CLINICAL TRIAL: NCT02655380
Title: Remifentanil Requirement for Acceptable Intubating Condition With Two Dose Ketamine Without Neuromuscular Blocking Agent in Children
Brief Title: Remifentanil Requirement for Acceptable Intubating Condition
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, yun jeong chae, Associate Professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MED-DRU-15-354
Record Dates: First submitted 2016-01-08; First posted 2016-01-14 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Intubating Condition
MeSH Terms: interventions — Remifentanil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ketamine 1 (Experimental): Anesthesia induction with ketamine 1 mg followed by remifentanil.
  Interventions: Drug: Ketamine 1; Drug: Remifentanil
- ketamine 2 (Experimental): Anesthesia induction with ketamine 2 mg followed by remifentanil.
  Interventions: Drug: Ketamine 2; Drug: Remifentanil

INTERVENTIONS:
Drug: Ketamine 1 — Anesthesia induction is performed with 1 mg ketamine.
  Arms: ketamine 1
Drug: Ketamine 2 — Anesthesia induction is performed with 2 mg ketamine.
  Arms: ketamine 2
Drug: Remifentanil — After anesthesia induction with ketamine, predetermined remifentanil using Dixon's up and dowm method is administered.

SUMMARY:
Ketamine and opioid are known to improve the intubating condition, respectively. Combination of ketamine and opioid potentiate analgesic effect and give hemodynamic stability in complementary manner. Therefore, the combination use of ketamine and remifentanil could be useful for acceptable intubating condition in the general anesthesia without the use of neuromuscular blocking agent. Generally, induction dose of ketamine ranges between 1 and 2 mg. There was no report about the optimal dose of remifentanil with 1 or 2 mg ketamine induction dose for intubation without neuromuscular blocking agent. The investigators focus on remifentanil dose using Dixon's up and down method.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II
* Undergoing general anesthesia with endotracheal tube

Exclusion Criteria:

* Anticipated difficult airway
* Patient with upper respiratory infection within 14 days
* Asthma

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2017-06-19 (Actual); Primary Completion 2018-04-16 (Actual); Study Completion 2018-04-16 (Actual)

PRIMARY OUTCOMES:
acceptability of intubation condition | during and after intubation, about 2 minute
  For assessment of intubation condition, 5 variables will be individually evaluated though 3 point scale (excellent, good, poor). If all variables are graded as excellent, intubation condition will be excellent. If at least 1 variable is poor, it will be reported as poor. Otherwise, it will be reported as good. Good and excellent will be considered to be acceptable intubating condition. Poor will be reported as unacceptable intubating condition.
  1. Laryngoscope easiness
  2. Vocal cord position
  3. Vocal cord movement
  4. Movement of limb
  5. Coughing

CONTACTS AND LOCATIONS:
Overall Officials: yun jeong chae, Ph.D, Study Director — Ajou University School of Medicine
Locations (1):
- Ajou universitiy school of medicine, Suwon, Gyeong-gi Do, South Korea